CLINICAL TRIAL: NCT05868174
Title: A Phase 1b Dose Escalation/Expansion Study of the Combination of 177Lu-TLX250 and Peposertib in Patients With Carbonic Anhydrase IX (CAIX)-Expressing Solid Tumors
Brief Title: Combination of 177Lu-TLX250 and Peposertib in Patients With Carbonic Anhydrase IX -Expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-TLX250-001
Record Dates: First submitted 2023-04-24; First posted 2023-05-22 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor, Adult; Advanced Solid Tumor; Advanced Renal Cell Carcinoma
Keywords: CAIX
MeSH Terms: interventions — peposertib

STUDY DESIGN:
Intervention Model Description: Dose escalation/de-escalations will be supported by the guidance given by outputs of the Bayesian model-based dose-escalation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-TLX250, 177Lu-TLX250 and Peposertib (Experimental): Diagnostic test: A single IV administration of 37 Megabecquerel (+/- 10%) 89Zr-DFO-girentuximab, containing a mass dose of 10 mg of girentuximab, followed by a diagnostic scan
  Treatment test: A single IV administration that could be 1887 - 2516 or 3145 Megabecquerel (+/- 10%) 177Lu-DOTA-girentuximab,containing a mass dose of 10 mg of girentuximab, on Day 1 of each 84-day cycle and p.o. administration of that could be 100-150 or 200 mg Peposertib BID on days 4-21 of each 84-day cycle.
  Interventions: Diagnostic Test: 89Zr-TLX250; Combination Product: 177Lu-TLX250 and Peposertib

INTERVENTIONS:
Diagnostic Test: 89Zr-TLX250 — Single IV administration followed by 89Zr-DFO-girentuximab PET/CT (or PET/MRI) scan at screening and approximately 8-10 weeks (±1 week) after Cycle 3 Day 1, as well as at the end of treatment visit (if feasible). The PET/CT should be obtained within 4-7 days after 89Zr-TLX250 administration
  Other Names: 89Zr-DFO-girentuximab
Combination Product: 177Lu-TLX250 and Peposertib — Dose escalation and de-escalation for the determination of the Maximum tolerated combination/ Recommended phase 2 dose.
  All subjects will receive 177Lu-TLX250 intravenously on day 1 and Peposertib BID on days 4-21 of each 84-day cycle.
  Other Names: 177Lu-DOTA-girentuximab

SUMMARY:
This is an open label, single-arm, multicentre dose escalation (Part 1) and dose expansion (Part 2) study to evaluate different combinations of 3 radioactive dose levels of 177Lu-TLX250 administered intravenously with 3 different doses of peposertib in patients with CAIX-expressing solid tumors.

DETAILED DESCRIPTION:
Part 1 (dose escalation) will evaluate the combination of 3 different activities of 177Lu-TLX250 and 3 different dose levels of peposertib.

Patients with CAIX positive solid tumors will be enrolled in a given dose/activity level in Cohorts of approximately 2-6 patients.

Treatment cycles will have a fixed length of 84 days. Patients will be treated during 3 cycles, or until clinically significant progression or unacceptable toxicity.

Part 2 (dose expansion) patients will be enrolled in 2 Cohorts:

* Cohort A: 40 patients with metastatic or non-resectable ccRCC
* Cohort B: 20 patients with CAIX-positive solid tumors (excluding RCC).

Patients will be treated at the Recommended phase 2 dose of 177Lu-TLX250 in combination with peposertib at the dosing schedule of the selected Recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic solid tumor that has progressed on or during/after recognized standard of care therapies and are not eligible for resection, or patients that are not eligible or not consenting to recognized standard of care therapies.
* At least one measurable lesion on CT/MRI according to RECIST 1.1 with corresponding 89Zr-TLX250 uptake (i.e., CAIX positive).
* CAIX positivity in at least 75% of the total lesion volume (defined as 89Zr- TLX250 uptake with intensity significantly greater than normal liver [i.e., standardized uptake value [SUV]max at least 1.5 times SUV of normal liver]).
* ECOG status 0 or 1.
* Have adequate organ function during screening
* Must have a life expectancy of at least 6 months.

Exclusion Criteria:

* Prior 177Lu-TLX250 or other radioligand therapy; or any prior CAIX targeting therapy.
* Known hypersensitivity to compounds of similar chemical or biologic composition to peposertib, girentuximab radiolabelled by zirconium or lutetium, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
* Administration of any radionuclide within 10 half-lives of the radionuclide prior to signature of the ICF.
* Patients who have had chemotherapy, definitive radiation, biological cancer therapy, or investigational agent/device within 28 days of first planned dose of study therapy.
* Patients who had > 2 prior lines of cytotoxic chemotherapy or had Grade 4 neutropenia or Grade 3/Grade 4 thrombocytopenia (both of a duration of at least 48 hours) during the last line of therapy. Note: This criterion may be removed in total or in part by the SRC upon review of the safety data from the initial dose level(s).
* Patients who cannot discontinue concomitant medications or herbal supplements that are strong inhibitors or strong inducers of cytochrome P450 (CYP) isoenzymes CYP3A4/5, CYP2C9, and CYP2C19. Concomitant use of CYP3A4/5 substrates with a narrow therapeutic index are also excluded.
* Patients who cannot discontinue concomitant H2-blockers or proton-pump inhibitors (PPIs). Patients may confer with the investigator to determine if such medications can be discontinued. These must be discontinued ≥ 5 days prior to study treatment. Patients do not need to discontinue calcium carbonate.
* Patients who are receiving therapeutic doses of anticoagulation, including but not limited to low-molecular weight heparin in therapeutic dosing or platelet aggregation inhibitors. Note: This criterion may be removed by the SRC upon review of the safety data from the initial dose level(s).
* Patients with ≥ 5 bone metastases and/or bulky (> 3cm in diameter) pelvic or femoral tumors, and/or metastases/tumor in the vertebral spine involving > 3 vertebrae.
* Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
* Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Requirement of concurrent use of other anti-cancer treatments or agents other than study medications. Supportive care therapies are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety parameter Dose Limited Toxicity (DLT) | 42 days
  Dose level toxicity evaluation using Partial Ordering Bayesian Logistic Regression Model Method (PO-BLRM)
Safety parameter Laboratory Examinations | 42 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding Laboratory examinations
Safety parameter Vital signs | 42 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding the vital signs
Safety parameter ECG | 42 days
  Frequency of occurrence and severity of abnormal findings in the 12-lead ECG (ECG QT interval)
Safety parameter Adverse Events and Treatment-Related Adverse Events | 42 days
  Assessment of AEs graded by the Common Terminology Criteria for Adverse Events (CTCAE) Criteria, Version 5.0
Disease impact causing changes in Eastern Cooperative Oncology Group (ECOG) Performance scale. | Screening/Baseline, Day1, Day 29, D57 and End of Treatment
  Quality of life ( in terms of their ability to care for themself, daily activity, and physical ability (walking, working) is to be evaluated using the ECOG Performance Scale.

SECONDARY OUTCOMES:
Overall Survival (OS) | Every 3 months ± 2 weeks for 24 months after the last 177Lu-TLX250 administration
  Overall Survival (OS), determined from enrollment , until death from any cause
Tumor objective response rate (ORR) | Every 3 months ± 2 weeks for 12 months after the last 177Lu-TLX250 administration
  Tumor response in terms of objective response rate (ORR) (solid tumor tissue response and overall radiological response [tumor response by RECIST 1.1 and overall radiological response by RECIST 1.1])
Progression-free survival (PFS) | Every 3 months ± 2 weeks for 12 months after the last 177Lu-TLX250 administration
  Progression free survival (PFS) defined as the time from enrollment to disease progression confirmed by radiology, clinical progression or death (whichever comes first)
Immunogenicity by formation of ADA(HACA) in blood | 84 days
  This outcome will be measured by analyzing the incidence of ADA(HACA) formation in blood on day 1, day 22, Day 43, Day 57 of each cycle (each cycle is 84 days) and at the end of treatment visit.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Macquarie University, North Ryde, New South Wales
  - Ashford (Icon) Cancer Centre, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - Austin Health, Melbourne
  - GenesisCare Murdoch, Perth